CLINICAL TRIAL: NCT06332053
Title: A Randomized, Open-label, Two-period, Self-controlled Study to Evaluate the Effect of Oral Rifampicin or Itraconazole on the Pharmacokinetics of SY-5007 Tablets in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Itraconazole and Rifampicin on the Pharmacokinetics of SY-5007 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SY-5007-I-03
Record Dates: First submitted 2024-03-14; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Healthy Subjects
Keywords: SY-5007 tablets; Itraconazole; Rifampin; Drug-drug Interaction Study
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A, Treatment Sequence (SY-5007-SY-5007/Itraconazole) (Experimental): SY-5007 80mg, tablets, once daily on Day 1 and Day 11 before meal; Itraconazole 200mg, once or twice daily from Day 8 to Day 18.
  Interventions: Drug: SY-5007; Drug: Itraconazole
- Group B, Treatment Sequence (SY-5007-SY-5007/Rifampin) (Experimental): SY-5007 160mg, tablets, once daily on Day 1 and Day 16 before meal, Rifampicin 600mg, once daily from Day 8 to Day 21.
  Interventions: Drug: SY-5007; Drug: Rifampin

INTERVENTIONS:
Drug: SY-5007 — SY-5007 80 mg, Tablets, 2 discrete single doses at Day 1 and Day 11
  Arms: Group A, Treatment Sequence (SY-5007-SY-5007/Itraconazole)
Drug: Itraconazole — Itraconazole 200 mg, Capsules, Day 8-Day 18
  Arms: Group A, Treatment Sequence (SY-5007-SY-5007/Itraconazole)
Drug: SY-5007 — SY-5007 160 mg, Tablets, 2 discrete single doses at Day 1 and Day 16
  Arms: Group B, Treatment Sequence (SY-5007-SY-5007/Rifampin)
Drug: Rifampin — Rifampin 600 mg, Capsules, Day 8-Day 21
  Arms: Group B, Treatment Sequence (SY-5007-SY-5007/Rifampin)

SUMMARY:
This study is a single-center, open-lable and fixed sequence test conducted in healthy subjects to evaluate the pharmacokinetic effects of Itraconazole and Rifampicin on a single dose of SY-5007 Oral administration. It is planned to enroll 28 healthy subjects and assign them to two parallel test groups, Group A (SY-5007 combined with Itraconazole) and Group B (SY-5007 combined with Rifampicin).

DETAILED DESCRIPTION:
A total of 28 evaluable healthy male subjects will be enrolled in this study. The subjects will be divided into two groups, A and B, with 14 people in each group.

In the itraconazole study (Group A), patients received single-dose SY-5007 80 mg on Day 1 and Day 11 and itraconazole 200 mg once or twice daily on Day 8-Day 18 orally.

In the rifampicin study (Group B), patients received single-dose SY-5007 160mg on Day 1 and Day 16 and rifampicin 600 mg once daily on Day 8-Day 21 orally.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Fully understand the purpose, nature, methods, and potential adverse reactions of the trial, voluntarily participate, and sign a written informed consent form (ICF), and be able to follow the protocol requirements to complete the study as healthy subjects.
2. Male subjects aged ≥18 and ≤45 years old (including boundary values, based on the time of signing the informed consent form).
3. Body weight ≥50kg, and body mass index (BMI = weight/height^2, kg/m^2) between 18 and 26 kg/m^2 (including boundary values).
4. Qualified subjects of reproductive capability must agree with their sexual partners to adopt a medically accepted contraceptive measure (such as intrauterine device, contraceptive pills, or condoms) during the trial and for 3 months after the end of the trial, and have no plans to donate sperm/eggs during the trial and for 3 months after the end of the trial.

Exclusion Criteria:

Subjects will be ineligible for this study if they meet any of the following criteria:

1. Clear history of severe allergies, non-allergic drug reactions, or multiple drug allergies, or known hypersensitivity reactions to the investigational drug (active pharmaceutical ingredient or excipients).
2. Positive for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen, hepatitis C antibodies, or syphilis treponema antibodies at screening.
3. Presence of clinically significant abnormal vital signs, physical examination findings, laboratory test results, or electrocardiogram results at screening.
4. Currently suffering from or known by the investigator to have chronic gastrointestinal, liver, or kidney diseases that may affect trial outcomes.
5. Symptoms or medical history of any major diseases, including but not limited to cardiovascular, hepatic, renal diseases, or other acute or chronic gastrointestinal diseases, respiratory diseases, musculoskeletal diseases, as well as diseases of the blood, endocrine, nervous, or psychiatric systems, or any other conditions or physiological states that may interfere with trial results.
6. Any surgical conditions or conditions that may significantly affect drug absorption, distribution, metabolism, and excretion, or any surgical conditions or conditions that may pose harm to subjects participating in the trial, such as a history of gastrointestinal surgery (gastrectomy, gastrojejunal anastomosis, intestinal resection, etc.), urinary tract obstruction or difficulty in urination, history of digestive tract ulcers, gastrointestinal bleeding, etc. (Subjects who have undergone appendectomy or hernia repair surgery can be enrolled in the study).
7. Known or suspected history of drug abuse within the past two years at screening, or drug abuse within the past three months at screening or baseline, or positive drug abuse screening during screening or baseline.
8. Underwent major surgery within the past six months before the first dose or planning to undergo surgery during the trial.
9. Smoked an average of more than 5 cigarettes per day within the past three months before the first dose or unwilling to stop using any tobacco products during the trial.
10. Regularly consumed alcohol within the past three months before the first dose (defined as consuming more than 14 units of alcohol per week, with 1 unit equal to 360 mL of beer with an alcohol content of 5%, or 45 mL of spirits with an alcohol content of 40%, or 150 mL of wine with an alcohol content of 12%), or unable to stop drinking during the trial, or positive alcohol breath test at screening.
11. History of blood donation or significant blood loss (≥300 mL) within the past two years before the first dose, or use of blood products or receiving blood transfusions within the past month before the first dose.
12. Participated in other drug or medical device clinical trials within the past three months before the first dose (excluding those screened but ultimately not enrolled), or used the study drug before.
13. Received vaccination or inactivated vaccines within the past month before the first dose.
14. Used any prescription drugs, non-prescription drugs, health products, or herbal medicines within the past two weeks before the first dose (if the half-life (t1/2) of the drug used can be confirmed, the washout period should be ≥5 t1/2, with the longer one taken).
15. Habitually consumed grapefruit juice or excessive amounts (more than 8 cups, 1 cup = 250 mL) of tea, coffee, and/or caffeinated beverages and unable to stop drinking for at least 48 hours before the first dose and during the trial.
16. Have special dietary requirements or difficulty swallowing.
17. Difficulty in blood sampling, or a history of fainting or intolerance to venipuncture.
18. Clear history of neurological or psychiatric disorders, including dementia or epilepsy, etc.
19. Diagnosis of malignant tumors within the past five years (excluding cured in situ cancers, such as non-melanoma skin cancers).
20. For scientific reasons, compliance reasons, or for the safety of the subjects, the investigator deems it inappropriate for the subject to participate in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Cmax for SY-5007 | Day 1-Day 22
  Defined as maximum observed plasma concentration
Tmax for SY-5007 | Day 1-Day 22
  Defined as time to maximum plasma concentration
AUC0-t for SY-5007 | Day 1-Day 22
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration
AUC0-∞ for SY-5007 | Day 1-Day 22
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to infinity
t½ for SY-5007 | Day 1-Day 22
  Defined as apparent plasma terminal phase disposition half-life
CL/F for SY-5007 | Day 1-Day 22
  Defined as apparent total body clearance
Vz/F for SY-5007 | Day 1-Day 22
  Defined as apparent oral Volume of distribution

SECONDARY OUTCOMES:
Safety of SY-5007 | Up to 29 days
  AE (adverse event) will be summarized by type and severity

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China